CLINICAL TRIAL: NCT06991933
Title: Preparation and Construction of Volumetric Plastination Models of the Limbic System, Basal Nuclei, Cerebellum, and Human Spinal Cord and Evaluation of Their Educational Effects
Brief Title: Construction and Educational Impact of Plastination Models of the Limbic System, Basal Nuclei, Cerebellum, and Human Spinal Cord
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, mehrnoush malekzadeh, Assistant Professor, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IR.ARI.MUI.REC.1404.007; 1403315 (Other Grant/Funding Number: Isfahan university medical sciences)
Record Dates: First submitted 2025-05-10; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Education; Education, Medical; Education, Medical, Undergraduate
Keywords: Medical education; Neuroanatomy; plastination model

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 : Plastination Model Group (Experimental): Receives instruction using plastinated models of:
  * Brainstem
  * Limbic system
  * Basal ganglia
  * Cerebellum
  * Spinal cord
  Duration: 7 weeks of training (2 hours/week)
  Taught by professor who every year teaches neuroanatomy
  Assessment: Standardized anatomy exams + spatial reasoning tests
  Interventions: Behavioral: Plastination Model Group
- Traditional Methods Group (Active Comparator): Receives equivalent instruction using:
  * Standard textbook and 2D atlases (e.g., Netter's)
  * Lectures with 2D projections
  Matched in duration and instructor expertise
  Same assessment protocol as an experimental group
  Interventions: Behavioral: Traditional Methods Group

INTERVENTIONS:
Behavioral: Plastination Model Group — Model Specifications:
  "S10 silicone plastination models of brainstem structures (1:1 scale) with:
  • Sectioned at 2mm intervals to reveal internal architecture
  Arms: Arm 1 : Plastination Model Group
Behavioral: Traditional Methods Group — 1. Netter's Atlas of Human Anatomy (9th ed.)
  2. Standardized PowerPoint lectures
  Arms: Traditional Methods Group

SUMMARY:
Purpose:

This educational trial aims to assess whether plastination models for neuroanatomy training (limbic system, basal ganglia, cerebellum, spinal cord)" improve medical students' understanding of central nervous system anatomy compared to traditional educational methods. It will also evaluate student satisfaction with this teaching tool.

Key Questions:

1. Do plastination models for neuroanatomy training (limbic system, basal ganglia, cerebellum, spinal cord) enhance test scores in neuroanatomy examinations?
2. How do students perceive the educational value of these models?

Study Design:

Researchers will compare two teaching methods:

* Intervention group: Learns using plastination models for neuroanatomy training (limbic system, basal ganglia, cerebellum, spinal cord)
* Control group: Learns using standard 2D atlases, power point and plastic models

Participants will:

1. Complete a pre-intervention anatomy knowledge test
2. Attend 4 weekly neuroanatomy sessions using their assigned method
3. Take a post-intervention exam and satisfaction survey
4. Participate in focus groups about their learning experience

ELIGIBILITY:
Inclusion Criteria:

* Medical students in their third semester of training
* Currently enrolled in neuroanatomy coursework at Isfahan University of Medical Sciences
* No prior formal training with plastinated models
* Willing to attend all study sessions for 7 weeks
* Able to complete assessments in persian

Exclusion Criteria:

* Prior experience with plastinated models
* Currently taking neuroanatomy remediation courses
* Planned absences during >20% of study sessions

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-23 (Estimated); Primary Completion 2025-12-29 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Change in neuroanatomy knowledge scores assessed by the "Neuroanatomy Knowledge Assessment Test | Baseline, Week 4 post-intervention
  Scale Title: Neuroanatomy Knowledge Assessment Test (NKAT). Score Range: 0 (no correct answers) to 15 (all answers correct). Interpretation: Higher scores indicate better neuroanatomy knowledge (better outcome).

SECONDARY OUTCOMES:
Spatial understanding assessment | Post-intervention only
  Method: 3D spatial reasoning test (modified Vandenberg scale)
  Scoring: 1-5 Likert scale for structure identification accuracy
Student satisfaction assessed by the 10-item Student Satisfaction Survey (SSS) | Immediately after the intervention (Day 1)
  * Score Range: 1 (strongly disagree) to 5 (strongly agree).
  * Interpretation: Higher scores indicate greater satisfaction (better outcome).

IPD SHARING:
Plan to Share IPD: No